CLINICAL TRIAL: NCT03662178
Title: Investigating the Structured Use of Ultrasound Scanning for Fetal Growth (Oxford Growth Restriction Identification Programme (OxGRIP)) on Risk Factors for and the Incidences of Adverse Maternal, Fetal and Neonatal Outcome
Brief Title: Investigating the Structured Use of Ultrasound Scanning for Fetal Growth
Acronym: OxGRIP
Status: Recruiting | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Lawrence Impey, Principal Investigator, Oxford University Hospitals NHS Trust
Other Study IDs: 17/SC/0374
Record Dates: First submitted 2017-11-16; First posted 2018-09-07 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Stillbirth; Fetal Death; Fetal Growth Retardation; Small for Gestational Age; Fetal Growth Restriction; Perinatal Death; Intrauterine Growth Restriction
MeSH Terms: conditions — Stillbirth; Fetal Death; Fetal Growth Retardation; Perinatal Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fetal growth restriction during pregnancy represents one of the biggest risk factors for stillbirth (Gardosi et al, 2013), with 'about one in three term, normally formed antepartum stillbirths are related to abnormalities of fetal growth' (MBRRACE, 2015).

Therefore, antenatal detection of growth restricted babies is vital in order to be able to monitor and decide the appropriate delivery timing.

However, antenatal detection of SGA babies has been poor, varying greatly across trusts in England in those that calculate their rates (NHS England, 2016). Most trusts do not calculate their detection rates and rates are therefore unknown. It is estimated that routine NHS care detects only 1 in 4 growth restricted babies (Smith, 2015).

Oxford University Hospitals NHS Foundation Trust, in partnership with the Oxford Academic Health Science Network (AHSN) has introduced a clinical care pathway (the Oxford Growth Restriction Pathway (OxGRIP)) designed to increase the rates of detection of these at risk babies. The pathway is intended to increase the identification of babies who are at risk of stillbirth, in order to try to prevent this outcome, whilst making best usage of resources, and restricting inequitable practice and unnecessary obstetric intervention.

It has been developed with reference to a body of research, however, the individual parts of care provided have not been put together in a pathway in this manner before. Therefore it is important to examine whether the pathway meets its goals of improving outcomes for babies in a 'real world' setting.

The principles of the pathway are

1. A universal routine scan at 36 weeks gestation.
2. Additional growth scans at 28 and 32 weeks gestation based on a simplified assessment of risk factors and universal uterine artery Doppler at 20 weeks gestation.
3. Assessment of further parameters other than estimated fetal weight associated with adverse perinatal outcome (eg growth velocity, umbilical artery Doppler and CPR).

The clinical data routinely collected as a result of the introduction of the pathway offers a valuable and unique resource in identifying and analysing in the effects of the pathway on its intended outcomes and also in investigating and analysing other maternal, fetal and neonatal complications and outcomes, establishing normal / reference ranges for ultrasound values.

DETAILED DESCRIPTION:
There is no requirement for patient participation in this study. All data collected and analysed is routinely collected clinical data.

ELIGIBILITY:
Inclusion Criteria:

• All pregnant women receiving antenatal care at the Oxford University Hospitals NHS Foundation Trust (OUHFT) from January 2013 to 31st December 2019 with no exclusion criteria

Exclusion Criteria:

* Women who have opted out of research related to pregnancy in this pregnancy whilst receiving care by the OUHFT.
* If intrapartum care takes place outside of the OUHFT.

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All pregnant women receiving antenatal care at the Oxford University Hospitals NHS Foundation Trust (OUHFT) from January 2013 to 31st December 2019
Sampling Method: Probability Sample
Enrollment: 56000 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Impact of OxGRIP on Perinatal mortality according to gestation | 4 yrs
  Mortality (stillbirth and neonatal death per 1000 pregnancies) in the period after birth) assessed in 2 years before the programme and compared with the 2 years after the programme started. Assessed for all pregnancies and for those reaching 35 weeks' gestation

SECONDARY OUTCOMES:
Impact of the OxGRIP Pathway on service: number of scans | 6 yrs
  Number of Ultrasound Scans (>24 weeks gestation) performed per pregnancy
Impact of the OxGRIP Pathway on service - Consultant time | 6 yrs
  Number of Consultant appointments
Impact of the OxGRIP Pathway on service - intrapartum interventions | 6 yrs
  Proportion of all birth delivered as emergency and elective cesarean sections and instrumental deliveries
Risk Factors for adverse outcomes - ultrasound head circumference | 4 yrs
  Routinely collected ultrasound fetal measurements - Head Circumference. Physiological parameter
Risk Factors for adverse outcomes - ultrasound abdomen circumference | 4 yrs
  Routinely collected ultrasound fetal measurements - Abdominal Circumference.Physiological parameter
Risk Factors for adverse outcomes - ultrasound femur length | 4 yrs
  Routinely collected ultrasound fetal measurements - Femur Length. Physiological parameter
Risk Factors for adverse outcomes - ultrasound presentation | 4 yrs
  Fetal presentation at last scan before birth. Physiological parameter
Risk Factors for adverse outcomes - Doppler ultrasound | 4 yrs
  Uterine/umbilical artery/ middle cerebral artery Doppler values. Physiological parameter
Clinical outcomes during pregnancy and postnatal/neonatal period: hypertension | 4 yrs
  Diagnosis of pre eclampsia and related complications. Physiological parameter
Clinical outcomes during pregnancy and postnatal/neonatal period: diabetes | 4 yrs
  Diagnosis of Gestational Diabetes. Physiological parameter
Clinical outcomes during pregnancy and postnatal/neonatal period: mode of birth | 4 yrs
  Mode of Delivery
Clinical outcomes during pregnancy and postnatal/neonatal period: preterm birth | 4 yrs
  Number of preterm births by gestation per 1000 pregnancies
Clinical outcomes during pregnancy and postnatal/neonatal period: stillbirth | 4 yrs
  Antenatal fetal loss rate per 1000 pregnancies
Clinical outcomes during pregnancy and postnatal/neonatal period: intrapartum stillbirth | 4 yrs
  Intrapartum fetal loss rate per 1000 pregnancies
Clinical outcomes during pregnancy and postnatal/neonatal period: neonatal death | 4 yrs
  Neonatal death <30 days of age: rate per 1000 livebirths
Clinical outcomes during pregnancy and postnatal/neonatal period: infant | 4 yrs
  Neonatal/infant death >30 days of age <1year of age: per 1000 live births
Clinical outcomes during pregnancy and postnatal/neonatal period: neonatal admission | 4 yrs
  Adverse neonatal outcome - planned/unplanned admission to NICU: rate per 1000 pregnancies
Clinical outcomes during pregnancy and postnatal/neonatal period: HIE | 4 yrs
  Adverse neonatal outcome - diagnosis of HIE rate per 1000 pregnancies
Clinical outcomes during pregnancy and postnatal/neonatal period: cord gas | 4 yrs
  Cord Blood Gases outside normal range (umbilical cord arterial pH at birth <7.00 and <7.05)
Clinical outcomes during pregnancy and postnatal/neonatal period: Apgar | 4 yrs
  Apgar score at birth (continuous variable and rate of <7 at 5 mins)
Clinical outcomes during pregnancy and postnatal/neonatal period: size | 4 yrs
  Small for Gestational Age birthweight - by Hadlock and Intergrowth centiles. Physiological parameter
Normal ranges of antenatal ultrasound markers. | 4 yrs
  Development of normal range of routinely collected ultrasound measurements. Physiological parameter
Normal ranges of intrapartum markers. | 4 yrs
  Cardiotocograph results ( Dawes Redman Criteria). Physiological parameter

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Impey, FRCOG, Study Director — Oxford University Hospitals NHS Trust
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Chauhan SP, Magann EF. Screening for fetal growth restriction. Clin Obstet Gynecol. 2006 Jun;49(2):284-94. doi: 10.1097/00003081-200606000-00010. PMID 16721107
- [Background] Gardosi J, Francis A. Adverse pregnancy outcome and association with small for gestational age birthweight by customized and population-based percentiles. Am J Obstet Gynecol. 2009 Jul;201(1):28.e1-8. doi: 10.1016/j.ajog.2009.04.034. PMID 19576372
- [Background] Sovio U, White IR, Dacey A, Pasupathy D, Smith GCS. Screening for fetal growth restriction with universal third trimester ultrasonography in nulliparous women in the Pregnancy Outcome Prediction (POP) study: a prospective cohort study. Lancet. 2015 Nov 21;386(10008):2089-2097. doi: 10.1016/S0140-6736(15)00131-2. Epub 2015 Sep 7. PMID 26360240
- [Background] Stacey T, Thompson JM, Mitchell EA, Zuccollo JM, Ekeroma AJ, McCowan LM. Antenatal care, identification of suboptimal fetal growth and risk of late stillbirth: findings from the Auckland Stillbirth Study. Aust N Z J Obstet Gynaecol. 2012 Jun;52(3):242-7. doi: 10.1111/j.1479-828X.2011.01406.x. Epub 2012 Jan 25. PMID 22276935
- [Background] Papageorghiou AT, Kennedy SH, Salomon LJ, Ohuma EO, Cheikh Ismail L, Barros FC, Lambert A, Carvalho M, Jaffer YA, Bertino E, Gravett MG, Altman DG, Purwar M, Noble JA, Pang R, Victora CG, Bhutta ZA, Villar J; International Fetal and Newborn Growth Consortium for the 21st Century (INTERGROWTH-21st). International standards for early fetal size and pregnancy dating based on ultrasound measurement of crown-rump length in the first trimester of pregnancy. Ultrasound Obstet Gynecol. 2014 Dec;44(6):641-8. doi: 10.1002/uog.13448. Epub 2014 Nov 2. PMID 25044000
- [Background] Gardosi J, Madurasinghe V, Williams M, Malik A, Francis A. Maternal and fetal risk factors for stillbirth: population based study. BMJ. 2013 Jan 24;346:f108. doi: 10.1136/bmj.f108. PMID 23349424